CLINICAL TRIAL: NCT05041881
Title: Long-term Comparative Analysis of Visual Outcomes and Patients Satisfaction With 3 Intraocular Lenses: Trifocal, Accommodating and Monofocal
Brief Title: Long-term Comparative Analysis of Visual Outcomes With 3 Intraocular Lenses: Monofocal, Trifocal and Accommodating
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Andrea Janekova, Principal Investigator, Faculty Hospital Kralovske Vinohrady
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRIMACO
Record Dates: First submitted 2021-09-08; First posted 2021-09-13 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Intraocular Lens
Keywords: trifocal lens; accommodating lens; monofocal lens; optical phenomena; glare

STUDY DESIGN:
Intervention Model Description: each group consist of patient receiving one type of intraocular lens- trifocal, accommodating or monofocal
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Trifocal IOL group (Active Comparator): Patients implanted during cataract or refractive surgery with trifocal lens, which allowed to see for far, intermediate and near distance, but due to optic design having unwanted effect like optical phenomena and lower contrast sensitivity
  Interventions: Device: Trifocal lens AT LISA TRI, Zeiss
- Accommodating IOL group (Active Comparator): Patients implanted during cataract or refractive surgery with accommodating lens, which allowed to see for far and should improve intermediate distance better than monofocal lens do.
  Interventions: Device: Accommodating Tetraflex HD lens, Lenstec inc.
- Monofocal IOL group (Active Comparator): Patients implanted during cataract or refractive surgery with standard monofocal lens, which allowed to see for far but patients do not experiences optical phenomena or low contrast sensitivity.
  Interventions: Device: Monofocal lens, Softec HD

INTERVENTIONS:
Device: Trifocal lens AT LISA TRI, Zeiss — lens is made of hydrophilic acrylic material with square edge technology and having diffractive optic design
  Arms: Trifocal IOL group
Device: Accommodating Tetraflex HD lens, Lenstec inc. — lens is made of hydrophilic acrylic material with square edge technology and having monofocal optic design
  Arms: Accommodating IOL group
Device: Monofocal lens, Softec HD — lens is made of hydrophilic acrylic material with square edge technology and having monofocal optic design
  Arms: Monofocal IOL group

SUMMARY:
To compare visual outcomes, contrast sensitivity, glare occurrence, incidence of posterior capsule opacification (PCO) and subjective satisfaction in patients implanted with trifocal, accommodating and monofocal lens in long term period.

DETAILED DESCRIPTION:
The goal of cataract surgery is to remove lens opacity and restore vision. Nowadays most of the patients wanted to be spectacle independent. The desire of visual acuity for all distances increases the popularity of multifocal and trifocal lenses. As these type of lenses are mostly based on diffractive structure, there could be occurrence of unwanted optical phenomena and lower contrast sensitivity. The effort is to produce intraocular lens (IOL) with good vision for all distances without these unwanted effects. Increasing daily task for intermediate distance led to the new category of IOLs- EDOF( extended depth of focus) IOLS, which are based mostly on diffractive profiles too, but should have less optical phenomena occurrence. To completely remove glare, halo and retain standard good contrast sensitivity enhance monofocal lenses were invented, mostly based on spherical aberrations, but not achieving as good intermediate vision as multifocal or EDOF lenses do. Accommodating lenses should provide better intermediate distance without unwanted optical effects on vision.

This study is retro-prospective, comparing 3 different lenses in long-term period. First group includes patients with trifocal lens allowing patients to see for all distances, second group includes patients with implanted accommodating lens which allows good distance and better intermediate distance than monofocal. Third group include patients with standard monofocal lens. Preoperative data were collected retrospectively and one prospective visit was scheduled in period 36- 48 months after the surgery. Study is conducted in 2 eye centers- one in Slovakia Trenčín, one in Prague, Czech Republic. The study was approved by the Ethic committee of faculty hospital Hradec Kralove (202103 P08). and will enrolled up 40 patients in each category.

ELIGIBILITY:
Inclusion Criteria:

* phacoemulsification with one of the 3 types of lens implantation before 36 to 48months
* no other ocular pathology affecting visual acuity
* able to maintain follow up visit

Exclusion Criteria:

* corneal opacities or irregularities
* amblyopia
* glaucoma with change in visual fields
* any other type of ocular surgery than phacoemulsification with primary lens implantation

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of visual acuity for distance between groups | 36-48 months after surgery
  uncorrected distance visual acuity (UDVA) corrected distance visual acuity (CDVA)
Comparison of visual acuity for intermediate between groups | 36-48 months after surgery
  Uncorrected intermediate visual acuity (UIVA) Distance corrected intermediate visual acuity (DCIVA)
Comparison of near visual acuity between group 1 (trifocal lens) and group 2 (accommodating lens) | 36-48 months after surgery
  uncorrected near visual acuity (UNVA)
Contrast sensitivity comparison between groups | 36-48 months after surgery
  Photopic contrast sensitivity with glare Mesopic contrast sensitivity with glare Mesopic contrast sensitivity without glare
Incidence of posterior capsule opacification (PCO) | 36-48 months after surgery
  Incidence of PCO and needed Nd YAG capsulotomy treatment in each group

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Janekova, MD, Principal Investigator — Faculty Hospital Kralovske Vinohrady
Locations (2):
- Eye Center Prague, Prague, Czech Republic, Czechia
- Eye Center Sokolik, Trenčín, Slovakia